CLINICAL TRIAL: NCT07034612
Title: Effect of Pulsatile and Non-Pulsatile Cardiopulmonary Bypass Flow on Choroidal Circulation in Diabetic and Non-Diabetic Patients
Brief Title: Choroidal Changes During Cardiopulmonary Bypass
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SamsunKVC OCT
Record Dates: First submitted 2025-06-14; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Retinopathy (DR); Cardiopulmonary Bypass; Retinal Vascular Diseases
Keywords: Diabetic Retinopathy; Cardiopulmonary Bypass; Pulsatile Flow
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Diabetic - Pulsatile Flow: Diabetic patients undergoing elective coronary artery bypass grafting (CABG) with pulsatile cardiopulmonary bypass (CPB) flow. Preoperative and postoperative 1st month OCTA measurements will be taken.
- Diabetic - Non-Pulsatile Flow: Diabetic patients undergoing elective CABG with non-pulsatile CPB flow. OCTA measurements preoperatively and at 1 month postoperatively.
- Non-Diabetic - Pulsatile Flow: Non-diabetic patients undergoing elective CABG with pulsatile CPB flow. OCTA measurements preoperatively and at 1 month postoperatively.
- Non-Diabetic - Non-Pulsatile Flow: Non-diabetic patients undergoing elective CABG with non-pulsatile CPB flow. OCTA measurements preoperatively and at 1 month postoperatively.

SUMMARY:
This prospective observational study investigates the impact of pulsatile versus non-pulsatile cardiopulmonary bypass (CPB) flow on choroidal circulation in diabetic and non-diabetic patients undergoing elective coronary artery bypass grafting (CABG). A total of 104 patients aged 30 to 70 years will be included, with balanced distribution between diabetic and non-diabetic groups. Optical coherence tomography angiography (OCTA) will be performed preoperatively and at 1 month postoperatively to assess changes in choroidal vascularity. The primary objective is to determine whether the type of CPB flow affects choroidal microcirculation, particularly in diabetic patients. The findings may support more individualized perfusion strategies in patients at risk of ocular microvascular impairment.

DETAILED DESCRIPTION:
This prospective observational study aims to investigate the effects of pulsatile and non-pulsatile cardiopulmonary bypass (CPB) flow types on choroidal and retinal microcirculation in diabetic and non-diabetic patients undergoing elective coronary artery bypass graft (CABG) surgery. Previous literature suggests that pulsatile perfusion may enhance end-organ perfusion, but data on ocular microvascular circulation remain scarce, especially in diabetic patients.

A total of 104 patients between the ages of 30 and 70 will be enrolled and divided into four groups based on diabetes status and CPB flow type. Optical coherence tomography angiography (OCTA) will be performed preoperatively and at 1 month postoperatively to measure the choroidal vascularity index (CVI) and other retinal microvascular parameters.The primary outcome is the change in CVI between baseline and 1-month follow-up. Secondary outcomes include retinal microvascular changes and comparative analyses between diabetic and non-diabetic groups.By evaluating the relationship between CPB flow type and ocular perfusion, particularly in patients with longstanding diabetes, this study may provide evidence to support individualized CPB strategies to minimize ocular microvascular compromise in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 30 and 70 years
2. Undergoing elective, first-time coronary artery bypass graft surgery (CABG)
3. Stable metabolic status
4. For diabetic group: history of diabetes mellitus for more than 10 years
5. No significant ocular media opacity (e.g., cataract or vitreous hemorrhage)
6. No tremor or condition interfering with OCTA imaging
7. Aortic cross-clamp time ≤ 120 minutes

Exclusion Criteria:

1. Age <30 or >70 years
2. Re-do or emergency cardiac surgery
3. Diabetes duration <10 years (for diabetic group)
4. Unstable metabolic state or active infection
5. Presence of significant cataract, vitreous hemorrhage, or tremor
6. Contraindications to OCTA imaging

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective coronary artery bypass grafting, including diabetic and non-diabetic individuals, recruited at a single center (Samsun Training and Research Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Choroidal Vascularity Index (CVI) from Baseline to 1-Month Postoperative | 1 month after surgery
  CVI will be calculated from OCTA images preoperatively and 1 month postoperatively. Mean change in CVI will be compared between pulsatile and non-pulsatile CPB groups.

SECONDARY OUTCOMES:
Change in Retinal Vascular Density (RVD) | 1 month after surgery
  RVD will be assessed by OCTA and measured as vessel density (%) at baseline and 1-month post-op, compared between study groups.
Change in Foveal Avascular Zone (FAZ) Area | 1 month after surgery
  FAZ area will be measured preoperatively and 1 month postoperatively using OCTA, and compared across study groups.
Comparison of CVI Change Between Diabetic and Non-Diabetic Patients | 1 month after surgery
  Subgroup analysis of CVI change will be performed to assess whether diabetes status affects choroidal perfusion response to CPB flow type.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsun University Faculty of Medicine, Samsun, Turkey (Türkiye)